CLINICAL TRIAL: NCT03561090
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Trial of Oral IW-3718 Administered to Patients With Gastroesophageal Reflux Disease While Receiving Proton Pump Inhibitors
Brief Title: A Trial of IW-3718 for 8 Weeks in Patients With Persistent Gastroesophageal Reflux Disease (GERD) Receiving Proton Pump Inhibitors (PPIs)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Parallel IW-3718 Phase III trial did not meet pre-specified criteria.
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C3718-301
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease; GERD; Proton Pump Inhibitors; IW-3718
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1500 mg IW-3718 BID + PPI (Experimental): Three 500 mg IW-3718 tablets administered twice daily (BID), immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before the morning meal each day.
  Interventions: Drug: IW-3718; Drug: Standard-dose PPIs QD
- Placebo + PPI (Placebo Comparator): Three placebo tablets administered BID immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before the morning meal each day.
  Interventions: Drug: placebo; Drug: Standard-dose PPIs QD

INTERVENTIONS:
Drug: IW-3718 — oral tablet
  Arms: 1500 mg IW-3718 BID + PPI
Drug: placebo — oral tablet
  Arms: Placebo + PPI
Drug: Standard-dose PPIs QD — background therapy

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of IW-3718 administered to patients with GERD who continue to have persistent symptoms, such as heartburn and regurgitation, while receiving once-daily (QD), standard-dose PPIs.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be eligible for enrollment in this study:

* Patient is an ambulatory male or female (if female, nonpregnant) and is at least 18 years old at the Screening Visit.
* Patient has a diagnosis of GERD and reports experiencing GERD symptoms (heartburn or regurgitation) while taking standard PPI therapy.
* Patient has evidence of pathological acid reflux.
* Female patients must not be pregnant and must agree to avoid pregnancy for the duration of the study.
* Patient must comply with study procedures.

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible to participate in the study:

* Patient has a history of complete lack of GERD symptom response to PPI therapy.
* Patient has a significant medical or surgical history including conditions that would impact drug absorption or metabolism (such as bowel obstruction, poorly controlled diabetes, gastroparesis, hiatal hernia).
* Patient reports pain or burning behind the breastbone or in the center of the upper stomach as his or her predominant symptom at the Screening Visit.
* Patient has received an investigational drug during the 30 days before the Screening Visit, or is planning to receive another investigational drug or use an investigational device at any time during the study.

NOTE: Other inclusion and exclusion criteria apply, per the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Shetzline, MD, PhD, Study Chair — Chief Medical Officer
Locations (99):
- United States (93):
  - Pinnacle Research Group, Anniston, Alabama
  - Alabama Medical Group, PC, Mobile, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Adobe Clinical Research LLC, Tucson, Arizona
  - Applied Research Center, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Anaheim Clinical Trials LLC - ERN-PPDS, Anaheim, California
  - GW Research, Inc., Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Facey Medical Foundation, Mission Hills, California
  - Northern California Research Corp, Sacramento, California
  - Digestive Care Center, San Carlos, California
  - Precision Research Institute, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Chase Medical Research LLC, Waterbury, Connecticut
  - West Central Gastroenterology, LLP, Clearwater, Florida
  - Avail Clinical Research LLC, DeLand, Florida
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - Borland Groover Clinic, Jacksonville, Florida
  - Health Awareness Inc - MRA, Jupiter, Florida
  - Millennium Clinical Research Inc-Miami, Miami, Florida
  - Advanced Research Institute, Inc, New Port Richey, Florida
  - Legacy Clinical Solutions: Sensible HealthCare, LLC - BTC - PPDS, Ocoee, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Pines Clinical Research Inc, Pembroke Pines, Florida
  - DMI Research, Pinellas Park, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Atlanta Center For Gastroenterology PC, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Avicenna-DM Clinical Research, Oak Lawn, Illinois
  - Iowa Digestive Disease Center, Clive, Iowa
  - West Glen GI, Shawnee Mission, Kansas
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - CroNOLA, LLC., Houma, Louisiana
  - Clinical Trials Management LLC, Mandeville, Louisiana
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Alan A Rosen MD PA, Baltimore, Maryland
  - Elligo Health Research, Frederick, Maryland
  - Meritus Center For Clinical Research, Hagerstown, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Clinical Research Professionals, Chesterfield, Missouri
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Advanced Research Institute - Reno, Reno, Nevada
  - AGA Clinical Research Associates, LLC. - MRA, Egg Harbor, New Jersey
  - Lovelace Scientific Resources Inc, Albuquerque, New Mexico
  - NYU School of Medicine, Great Neck, New York
  - Beth Israel Medical Center, New York, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Orchard Park Family Practice, Orchard Park, New York
  - Medication Management LLC, Greensboro, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - East Carolina Gastroenterology, Jacksonville, North Carolina
  - Wake Endoscopy Center, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Consultants For Clinical Research Inc, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Legacy Research Institute, Portland, Oregon
  - Veterans Research Foundation of Pittsburgh - NAVREF, Pittsburgh, Pennsylvania
  - Consultants of Gastroenterology, Columbia, South Carolina
  - WR - ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Multi Specialty Clinical Research, Johnson City, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Gastroenterology-Union City, Union City, Tennessee
  - Dallas VA Medical Center - NAVREF, Dallas, Texas
  - Digestive Health Associates of Texas, Garland, Texas
  - Biopharma Informatic Inc., Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Research Consultants, Houston, Texas
  - Houston Digestive Diseases Clinic, Houston, Texas
  - Pearland Physicians, Pearland, Texas
  - Quality Research Inc, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Advanced Research Institute, Ogden, Utah
  - Aspen Clinical Research LLC - MRA, Orem, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - GI Associates Gainesville, Gainesville, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Washington Gastroenterology, Bellevue, Washington
  - Mayo Clinic Health System - Franciscan Healthcare - PPDS, La Crosse, Wisconsin
  - Wisconsin Center for Advanced Research Division of GI Associates, Milwaukee, Wisconsin
- Canada (6):
  - ALTA Clinical Research Inc, Edmonton, Alberta
  - Taunton Surgical Centre, Oshawa, Ontario
  - Digestive Health Clinic, Richmond Hill, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Digestive Disease Associates Inc, Vaughan, Ontario
  - Recherche Clinique Sigma, Inc., Québec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the screening and pre-treatment periods, participants were stratified by whether they had/did not have erosive esophagitis (EE) on esophagogastroduodenoscopy (EGD), and by their baseline weekly heartburn severity score (WHSS, defined as the average heartburn severity score over the last 7 days prior to randomization of < 3 vs. ≥ 3), and were randomly assigned 1:1 within each stratum to placebo or 1500 mg IW-3718 twice daily (BID).
Groups:
- Placebo BID + PPI: Three placebo tablets administered BID immediately after the morning and evening meals. Standard-dose proton pump inhibitors (PPIs) administered QD approximately 30-60 minutes before the morning meal each day.
- 1500 mg IW-3718 BID + PPI: Three 500 mg IW-3718 tablets administered BID, immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before the morning meal each day.
Period: Overall Study
Arm/Group | Placebo BID + PPI | 1500 mg IW-3718 BID + PPI
Started (Randomized) | 247 | 248
Randomized and Treated | 246 | 247
Completed | 207 | 212
Not Completed | 40 | 36
Not completed — Adverse Event | 11 | 7
Not completed — Non-Compliance With Study Drug | 2 | 0
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Lost to Follow-up | 7 | 2
Not completed — Study Terminated by Sponsor | 10 | 15
Not completed — Randomized by Mistake | 1 | 1
Not completed — Other Not Specified | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population: randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo BID + PPI: Three placebo tablets administered BID immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before the morning meal each day.
- Total: Total of all reporting groups
Arm/Group | Placebo BID + PPI | 1500 mg IW-3718 BID + PPI | Total
Number analyzed (Participants) | 246 | 247 | 493
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.17) | 48.1 (12.61) | 47.6 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 145 | 309
  Male | 82 | 102 | 184
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 55 | 107
  Not Hispanic or Latino | 187 | 188 | 375
  Unknown or Not Reported | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 201 | 203 | 404
  Black or African American | 32 | 33 | 65
  Asian | 10 | 6 | 16
  Other, Not Specified | 3 | 5 | 8
Erosive Esophagitis (EE) Status, as Randomized [Count of Participants; unit: Participants] — Population: Modified Intent-to-Treat (mITT) Population, which included all participants who 1) were randomized prior to or on 04 August 2020, 2) had received at least 1 dose of study drug, and 3) had at least 1 postbaseline primary efficacy assessment.
  Participants
    EE Present: number analyzed (Participants) | 228 | 227 | 455
    EE Present | 101 | 103 | 204
    EE Not Present: number analyzed (Participants) | 228 | 227 | 455
    EE Not Present | 127 | 124 | 251
Weekly Heartburn Severity Score (WHSS) Category, as Randomized [Count of Participants; unit: Participants] — WHSS=weekly average of Daily Heartburn Severity Score (DHSS). DHSS=the greater of the 2 items assessing heartburn severity (#1=Burning feeling behind the breastbone or in the center of the upper stomach; #2=Pain behind the breastbone or in the center of the upper stomach), where 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, and 5=Severe; higher scores indicate worse symptoms.
  Baseline is derived from the daily eDiary data collected in the pretreatment period, specifically the period of time from 7 days before randomization up to the time of randomization. Population: mITT Population, which included all participants who 1) were randomized prior to or on 04 August 2020, 2) had received at least 1 dose of study drug, and 3) had at least 1 postbaseline primary efficacy assessment.
  Participants
    WHSS Score >/= 3: number analyzed (Participants) | 228 | 227 | 455
    WHSS Score >/= 3 | 136 | 140 | 276
    WHSS Score < 3: number analyzed (Participants) | 228 | 227 | 455
    WHSS Score < 3 | 92 | 87 | 179
WHSS [Mean (Standard Deviation); unit: score on a scale] — WHSS=weekly average of Daily Heartburn Severity Score (DHSS). DHSS=the greater of the 2 items assessing heartburn severity (#1=Burning feeling behind the breastbone or in the center of the upper stomach; #2=Pain behind the breastbone or in the center of the upper stomach), where 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, and 5=Severe; higher scores indicate worse symptoms.
  Baseline is derived from the daily eDiary data collected in the pretreatment period, specifically the period of time from 7 days before randomization up to the time of randomization. Population: mITT Population: participants who were randomized prior to or on 04 August 2020, and who received at least 1 dose of study drug and had at least 1 postbaseline primary efficacy assessment.
  score on a scale
    number analyzed (Participants) | 228 | 227 | 455
    (all) | 3.17 (0.66) | 3.25 (0.79) | 3.21 (0.73)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in WHSS at Week 8
Description: The WHSS is defined as the weekly average of the DHSS. The DHSS for a day is the greater of the 2 items assessing heartburn severity (Item #1 "Burning feeling behind the breastbone or in the center of the upper stomach" and Item #2 "Pain behind the breastbone or in the center of the upper stomach"). The DHSS items are assessed on a 5-point ordinal scale, where 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, and 5=Severe; higher scores indicate worse symptoms. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 8
Population: mITT Population: participants who were randomized prior to or on 04 August 2020, and who received at least 1 dose of study drug and had at least 1 postbaseline primary efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo BID + PPI | 1500 mg IW-3718 BID + PPI
Number analyzed (Participants) | 228 | 227
score on a scale | -1.774 (0.082) | -1.719 (0.082)
Statistical Analysis 1: Comparison: Placebo BID + PPI vs 1500 mg IW-3718 BID + PPI; Treatment difference calculated as least squares mean (LSM) change from baseline at Week 8; IW-3718 - placebo based on an mixed models repeated measures (MMRM) model with week (categorical), treatment group, week-by-treatment group, and week-by-baseline value interactions, baseline esophagitis status (present vs. not present), and baseline WHSS (< 3 vs. ≥ 3) as fixed effect terms and baseline value as a covariate, with subject as a random effect. An unstructured covariance structure was used; Test type: Superiority; p = 0.6346, MMRM; Least squares (LS) mean difference = 0.055, 95% CI 2-sided [-0.172 to 0.281] — Treatment difference (IW-3718 - placebo)

2. Secondary Outcome: Change From Baseline in Weekly Regurgitation Frequency Score (WRFS) at Week 8
Description: The WRFS is defined as the average of available daily regurgitation frequency scores (DRFS) during a week. DRFS is defined as the maximum score of the 2 items measuring regurgitation from a particular day (Item #6 "Regurgitation [liquid or food moving upwards toward your throat or mouth]" and Item #7 "An acid or bitter taste in the mouth"). The DRFS items are assessed on a 4-point ordinal scale, where 0=Never, 1=Rarely, 2-Sometimes, 3=Often, and 4=Very Often; higher scores indicate worse symptoms. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo BID + PPI | 1500 mg IW-3718 BID + PPI
Number analyzed (Participants) | 228 | 227
score on a scale | -1.330 (0.067) | -1.294 (0.068)
Statistical Analysis 1: Comparison: Placebo BID + PPI vs 1500 mg IW-3718 BID + PPI; Treatment difference calculated as LSM change from baseline at Week 8; IW-3718 - placebo based on an MMRM model with week (categorical), treatment group, week-by-treatment group, and week-by-baseline value interactions, baseline esophagitis status (present vs. not present), and baseline WHSS (< 3 vs. ≥ 3) as fixed effect terms and baseline value as a covariate, with subject as a random effect. An unstructured covariance structure was used; Test type: Superiority; p = 0.7101, MMRM; LS Mean Difference = 0.035, 95% CI 2-sided [-0.151 to 0.221] — Treatment difference (IW-3718 - placebo)

3. Secondary Outcome: Percentage of Participants Who Were Overall Heartburn Responders During the 8-Week Treatment Period
Description: An overall heartburn responder is a participant who is a weekly heartburn responder for at least 4 of the 8 treatment weeks and for at least 1 of the final 2 treatment weeks (i.e., Week 7 and Week 8). A weekly heartburn responder is a participant with a decrease of >/= 45% from baseline in WHSS. A participant who reported heartburn severity for less than 4 days during a week is not considered a responder for that week.
  The WHSS is defined as the weekly average of the DHSS. The DHSS for a day is the greater of the 2 items assessing heartburn severity (Item #1 "Burning feeling behind the breastbone or in the center of the upper stomach" and Item #2 "Pain behind the breastbone or in the center of the upper stomach"). The DHSS items are assessed on a 5-point ordinal scale, where 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, and 5=Severe; higher scores indicate worse symptoms. A negative change from baseline indicates improvement
Time Frame: Up to Week 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo BID + PPI | 1500 mg IW-3718 BID + PPI
Number analyzed (Participants) | 228 | 227
percentage of participants | 53.1 [46.4 to 59.7] | 47.6 [40.9 to 54.3]
Statistical Analysis 1: Comparison: Placebo BID + PPI vs 1500 mg IW-3718 BID + PPI; Test type: Superiority; Difference in percentage of responders = -5.5, 95% CI 2-sided [-14.7 to 3.7] — 95% confidence interval (CI) for Difference in Responder Rates is obtained using the Newcombe CI
Statistical Analysis 2: Comparison: Placebo BID + PPI vs 1500 mg IW-3718 BID + PPI; Treatment difference was calculated as the difference in the responder rates at Week 8; IW-3718 - placebo. The 95% CI for the difference in the responder rates was obtained using the Newcombe CI. P value was based on the odds ratio for the response rate (IW-3718:placebo) obtained from the CMH tests controlling for baseline esophagitis status and baseline heartburn severity level (< 3 vs. ≥ 3); Test type: Superiority; p = 0.2531, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.56 to 1.17] — Odds Ratio for Response (IW-3718 : placebo)

4. Secondary Outcome: Proportion of Heartburn-Free Days During the 8-Week Treatment Period
Description: Proportion of heartburn-free days is calculated as the number of heartburn-free (DHSS=0) days divided by the number of diary entry days. The DHSS for a day is the greater of the 2 items assessing heartburn severity (Item #1 "Burning feeling behind the breastbone or in the center of the upper stomach" and Item #2 "Pain behind the breastbone or in the center of the upper stomach"). The DHSS items are assessed on a 5-point ordinal scale, where 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, and 5=Severe; higher scores indicate worse symptoms. A negative change from baseline indicates improvement
Time Frame: Up to Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: proportion of days
Groups:
- Placebo BID + PPI: Three placebo tablets administered BID, immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before the morning meal each day.
- 1500 mg IW-3718 BID + PPI: Three 1500 mg IW-3718 tablets administered BID immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before the morning meal each day.
Arm/Group | Placebo BID + PPI | 1500 mg IW-3718 BID + PPI
Number analyzed (Participants) | 228 | 227
proportion of days | 0.232 (0.032) | 0.218 (0.031)
Statistical Analysis 1: Comparison: Placebo BID + PPI vs 1500 mg IW-3718 BID + PPI; Poisson regression including the fixed categorical effect of treatment, the baseline esophagitis status (present vs. not present) and baseline WHSS (<3 vs. ≥3), the covariate of baseline proportion of heartburn-free days, and with the diary entry duration (in days) as a weight variable adjusted in the model was applied; Test type: Superiority; p = 0.7445, Negative binomial model — Negative binomial model was used to deal with data overdispersion; Proportion ratio = 0.938, 95% CI 2-sided [0.636 to 1.382] — Proportion Ratio (1500 mg IW-3718 BID + PPI: Placebo + PPI)
Statistical Analysis 2: Comparison: Placebo BID + PPI vs 1500 mg IW-3718 BID + PPI; [analysis description as in outcome 4, analysis 1]; Test type: Other — Negative binomial model was used to deal with data overdispersion; Difference in Proportion Ratio = -0.015, 95% CI 2-sided [-0.103 to 0.074] — Difference in Proportion Ratio, (1500 mg IW-3718 BID + PPI) - (Placebo + PPI)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of treatment (up to Week 8) plus 7 days.
Description: Safety Population: Participants who received at least 1 dose of study drug.
Arm/Group | Placebo BID + PPI | 1500 mg IW-3718 BID + PPI
All-Cause Mortality (participants affected / at risk) | 0/246 | 0/247
Serious Adverse Events (participants affected / at risk) | 0/246 | 3/247
Other Adverse Events (participants affected / at risk) | 37/246 | 37/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID + PPI (N=246) | 1500 mg IW-3718 BID + PPI (N=247)
Cholecystitis (Hepatobiliary disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID + PPI (N=246) | 1500 mg IW-3718 BID + PPI (N=247)
Flatulence (Gastrointestinal disorders) | 10 | 9
Diarrhoea (Gastrointestinal disorders) | 17 | 8
Constipation (Gastrointestinal disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 6 | 6
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 8
Nasopharyngitis (Infections and infestations) | 2 | 5
Urinary tract infection (Infections and infestations) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT03561090/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT03561090/SAP_001.pdf